CLINICAL TRIAL: NCT05593328
Title: A Phase 2, Randomized, Open-label Study of Onvansertib in Combination With FOLFIRI and Bevacizumab Versus FOLFIRI and Bevacizumab for Second Line Treatment of Metastatic Colorectal Cancer in Patients With a KRAS or NRAS Mutation
Brief Title: Study of Onvansertib in Combination With FOLFIRI and Bevacizumab Versus FOLFIRI and Bevacizumab for Second Line Treatment of Metastatic Colorectal Cancer in Participants With a Kirsten Rat Sarcoma Virus Gene (KRAS) or Neuroblastoma-RAS (NRAS) Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cardiff Oncology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRDF-003
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Cancer; Metastatic Colorectal Cancer
Keywords: Colorectal Cancer; Metastatic Colorectal Cancer; KRAS Mutation; NRAS Mutation; Onvansertib; FOLFIRI; Bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — onvansertib; IFL protocol; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Onvansertib 20 mg + Standard of Care (SOC) (Experimental): Participants will receive 20 mg of onvansertib on Days 1 to 5 and 15 to 19 of a 28-day treatment cycle and SOC (FOLFIRI + bevacizumab) on Days 1 and 15 of each 28-day cycle.
  Interventions: Drug: Onvansertib; Drug: FOLFIRI; Drug: Bevacizumab
- Onvansertib 30 mg + Standard of Care (SOC) (Experimental): Participants will receive 30 mg of onvansertib on Days 1 to 5 and 15 to 19 of a 28-day treatment cycle and SOC (FOLFIRI + bevacizumab) on Days 1 and 15 of each 28-day cycle.
  Interventions: Drug: Onvansertib; Drug: FOLFIRI; Drug: Bevacizumab
- Standard of Care (SOC) (Active Comparator): Participants will receive SOC (FOLFIRI + bevacizumab) on Days 1 and 15 of each 28-day cycle.
  Interventions: Drug: FOLFIRI; Drug: Bevacizumab

INTERVENTIONS:
Drug: Onvansertib — Oral capsule
  Arms: Onvansertib 20 mg + Standard of Care (SOC); Onvansertib 30 mg + Standard of Care (SOC)
Drug: FOLFIRI — FOLFIRI (irinotecan + fluorouracil [5-FU] + leucovorin) as intravenous (IV) infusion
Drug: Bevacizumab — IV infusion

SUMMARY:
The primary objective of this study is to assess the efficacy of 2 different doses of onvansertib in combination with a chemotherapy regimen of irinotecan, fluorouracil [5-FU], and leucovorin (FOLFIRI) and bevacizumab for treatment of confirmed metastatic and/or unresectable colorectal cancer (CRC) in participants with a kirsten rat sarcoma virus gene (KRAS) or neuroblastoma-RAS (NRAS) mutation who have progressed on an oxaliplatin/fluoropyrimidinebased regimen in the first-line setting.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic and/or unresectable colorectal cancer (CRC).
2. Documentation of a kirsten rat sarcoma virus gene (KRAS) or neuroblastoma-RAS (NRAS) mutation in exon 2, 3, or 4 in primary tumor or metastasis, assessed by a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory.
3. Age ≥ 18 years.
4. Participants with tumors that have progressed on an oxaliplatin/fluoropyrimidine--based regimen with or without bevacizumab.

   1. Participants must have had systemic therapy within 180 days of the screening visit.
   2. Participants must have, at any time previously, received oxaliplatin-based chemotherapy with or without bevacizumab (≥ 6 weeks in duration).
   3. Participants who received oxaliplatin/fluoropyrimidine-based neoadjuvant, adjuvant, and/or fluoropyrimidine maintenance or adjuvant therapy and have disease recurrence or progression > 6 months from their last dose of oxaliplatin will be required to have received oxaliplatin/fluoropyrimidine-based therapy with or without bevacizumab as first-line treatment for metastatic disease.
   4. Participants who received an oxaliplatin-based regimen in the first-line setting and discontinued oxaliplatin because of toxicity or who received oxaliplatin for maintenance therapy are eligible as long as progression occurred < 6 months after the last dose of oxaliplatin therapy for advanced metastatic disease. It is recommended that these participants be re-challenged (if feasible) with oxaliplatin/fluoropyrimidine therapy and subsequently progress prior to eligibility. Participants with oxaliplatin-related neuropathy or oxaliplatin infusion-related hypersensitivity that cannot be rechallenged with oxaliplatin are eligible.
5. Participants must not have received prior treatment with irinotecan.
6. FOLFIRI therapy is appropriate for the participant as determined by the Investigator.
7. Imaging computed tomography (CT) or magnetic resonance imaging (MRI) of chest/abdomen/pelvis or other scans as necessary to document all sites of disease performed within 28 days prior to the first dose of onvansertib. Only participants with measurable disease as defined per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) are eligible for enrollment. CT is the preferred imaging modality, but MRI is also accepted. All subsequent scans must consistently use the same imaging modality for comparison with the Screening scan throughout the study.
8. Must have acceptable organ function
9. Signed informed consent to provide blood sample(s) for specific correlative assays

Exclusion Criteria:

1. Concomitant KRAS or NRAS and BRAF-V600 mutation or Microsatellite Instability High/Deficient Mismatch Repair (MSI-H/dMMR).
2. Anti-cancer chemotherapy or biologic therapy administered within 28 days prior to the first dose of study drug. The exception is a single dose of radiation up to 8 Gray (equal to 800 RAD) with palliative intent for pain control up to 14 days before enrollment, provided it is not the target lesion.
3. More than 1 prior chemotherapy regimen administered in the metastatic setting.
4. Major surgery within 6 weeks prior to enrollment.
5. Untreated or symptomatic brain metastasis.
6. Gastrointestinal (GI) disorder(s) that, in the opinion of the Investigator, would significantly impede the absorption of an oral agent (e.g., intestinal occlusion, active Crohn's disease, ulcerative colitis, extensive gastric and small intestine resection).
7. Unable or unwilling to swallow study drug.
8. Known hypersensitivity to fluoropyrimidine or leucovorin.
9. Known hypersensitivity to irinotecan.
10. Abnormal glucuronidation of bilirubin; known Gilbert's syndrome.
11. QT interval:

    1. Fridericia's correction (QTcF) > 470 milliseconds. The QTcF should be calculated as the arithmetic mean of the QTcF on triplicate electrocardiograms (ECGs). In the case of potentially correctible causes of QT prolongation that are readily corrected (e.g., medications, hypokalemia), the triplicate ECG may be repeated once during Screening and that result may be used to determine eligibility.
    2. Planned concomitant use of medications known to prolong the QT/QTc interval according to institutional guidelines.
    3. Presence of risk factors for torsade de pointes, including family history of Long QT Syndrome or uncorrected hypokalemia.
12. Use of strong cytochrome P450 3A4 (CYP3A4) or cytochrome P450 2C19 (CYP2C19) inhibitors or strong CYP3A4 inducers. Participants currently receiving these agents who can be switched to alternate therapy are not excluded. Inhibitors should be stopped at least 1 week prior to the first dose of protocol therapy and inducers should be stopped at least 2 weeks prior to initiation of protocol therapy.
13. The following are exclusion criteria for bevacizumab:

    1. History of cardiac disease: Congestive heart failure (CHF) Class II or higher according to the New York Heart Association (NYHA); active coronary artery disease, myocardial infarction within 6 months prior to study entry; unevaluated new onset angina within 3 months or unstable angina (angina symptoms at rest) or cardiac arrhythmias requiring anti-arrhythmic therapy, with the exception of participants who have been receiving therapy and are deemed by the Investigator to have stable/controlled disease.
    2. Current uncontrolled hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >90 mmHg despite optimal medical management) and prior history of hypertensive crisis or hypertensive encephalopathy.
    3. History of arterial thrombotic or embolic events (within 6 months prior to study entry).
    4. Significant vascular disease (eg, aortic aneurysm, aortic dissection, symptomatic peripheral vascular disease).
    5. Evidence of bleeding diathesis or clinically significant coagulopathy.
    6. Major surgical procedure (including open biopsy, significant traumatic injury, etc) within 28 days, or anticipation of the need for major surgical procedure during the study, and minor surgical procedure (excluding placement of a vascular access device) within 7 days prior to study enrollment.
    7. Proteinuria at Screening as demonstrated by urinalysis with proteinuria ≥2+ (participants discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate ≤1 g of protein in 24 hours to be eligible).
    8. Abdominal fistula, gastrointestinal perforation, peptic ulcer, or intra-abdominal abscess within the past 6 months.
    9. Ongoing serious, non-healing wound, ulcer, or bone fracture
    10. Known hypersensitivity to any component of bevacizumab
    11. History of reversible posterior leukoencephalopathy syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-03-17 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Up to approximately 1 year
  Defined as complete response (CR) or partial response (PR) as determined according to the Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) by an independent central review.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Up to approximately 1 year
  Defined from the date of first drug administration to progression or death, whichever occurs first.
Number of Participants with an Adverse Event (AE) | Up to approximately 1 year
  Type, incidence, causality and severity of AEs based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0. Clinically significant changes from baseline in vital signs, laboratory parameters, electrocardiograms (ECGs), physical examinations, weight, and Eastern Cooperative Oncology Group (ECOG) performance status will be recorded as AEs.
Disease Control Rate (DCR) | Up to approximately 1 year
  Defined as CR plus PR plus stable disease (SD).
Duration of Response (DOR) | Up to approximately 1 year
  Defined from the date of first response (CR or PR) to disease progression (PD) or death, whichever occurs first.
Overall Survival (OS) | Up to approximately 1 year
  Defined as the time from drug administration to death due to any cause.
Overall Response (OR) | Up to approximately 1 year
  Defined as CR or PR, PFS, DCR, DOR, and OS associated with a reduction in mutation allele frequency (MAF).
Maximum Concentration (Cmax) of Onvansertib | Day 1 and Day 5 of Cycle 1, and Day 5 of Cycle 3 (cycle is 28 days)
Area Under The Plasma Concentration Curve (AUC) of Onvansertib | Day 1 and Day 5 of Cycle 1, and Day 5 of Cycle 3 (cycle is 28 days)
Trough Concentration (Ctrough) of Onvansertib | Day 1 and Day 5 of Cycle 1, and Day 5 of Cycle 3 (cycle is 28 days)
Maximum Concentration (Cmax) of Onvansertib Metabolites | Day 1 and Day 5 of Cycle 1, and Day 5 of Cycle 3 (cycle is 28 days)
Area Under The Plasma Concentration Curve (AUC) of Onvansertib Metabolites | Day 1 and Day 5 of Cycle 1, and Day 5 of Cycle 3 (cycle is 28 days)
Trough Concentration (Ctrough) of Onvansertib Metabolites | Day 1 and Day 5 of Cycle 1, and Day 5 of Cycle 3 (cycle is 28 days)
Efficacy: Exposure Response Evaluation of Onvansertib | Up to approximately 1 year
  Correlation between onvansertib exposure and overall response rate.
Safety: Exposure Response Evaluation of Onvansertib | Up to approximately 1 year
  Correlation between onvansertib exposure and the number of participants with an AE.

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Mayo Clinic in Arizona - Phoenix Campus, Phoenix, Arizona
  - Central Arkansas Radiation Therapy Institute - Cancer Center, Little Rock, Arkansas
  - Pacific Cancer Medical Center, Anaheim, California
  - Comprehensive Blood and Cancer Center - Bakersfield, Bakersfield, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - Norris Comprehensive Cancer Center, Los Angeles, California
  - UCI Health - Chao Family Comprehensive Cancer Center, Orange, California
  - UCLA Health - Santa Monica Parkside Cancer Care, Santa Monica, California
  - Torrance Memorial Physician Network - Cancer Care and Infusion Center, Torrance, California
  - PIH Health, Whittier, California
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Cancer & Hematology Centers of Western Michigan - Lemmen-Holton Cancer Pavilion, Grand Rapids, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine Center for Advanced Medicine, St Louis, Missouri
  - Nebraska Cancer Specialists - Midwest Cancer Center - Legacy, Omaha, Nebraska
  - Englewood Health, Englewood, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - Manhattan Hematology Oncology Associates, New York, New York
  - Gabrail Cancer and Research Center, Canton, Ohio
  - Trihealth Kenwood, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - West Cancer Center - East Campus, Germantown, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - University of Virginia School of Medicine, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No